CLINICAL TRIAL: NCT02193490
Title: Safety and Efficacy Of Recombinant Human Deoxyribonuclease Eye Drops In Patients With Sjogren's and Non-Sjogren Dry Eye Disease
Brief Title: DNase Treatment for Dry Eyes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor ceased sponsorship and terminated the research citing slow accrual of subjects in this clinical trial.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Research to Prevent Blindness (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sandeep Jain, MD, Associate Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-1106
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye
Keywords: DNase, Pulmozyme, dry eye disease, treatment
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Deoxyribonucleases; dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DNase (Active Comparator): DNase 0.1% eye drops four times a day for 8 weeks
  Interventions: Drug: DNase
- Vehicle (Placebo Comparator): Drug vehicle eye drops four times a day for 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: DNase — DNase 0.1% eye drops four times a day for 8 weeks
  Other Names: Pulmozyme
  Arms: DNase
Drug: Vehicle — Drug vehicle eye drops four times a day for 8 weeks
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the tolerability and preliminary efficacy of DNase eye drops in patients with Sjogren's and Non-Sjogren Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Capable of giving informed consent and does provide informed consent.
* Documented Dry Eye Disease for at least 6 months.
* Schirmer I <10
* Corneal/ conjunctival (Rose Bengal) staining ≥1
* Ocular symptoms must be considered as annoying or activity limiting (OSDI ≥13; mild).
* Women must be post-menopausal ≥ 1 year, or surgically sterilized. If not, a negative urine pregnancy test is required within 14 days of receiving her first dose of test medication (placebo/ study drug) along with definite evidence of contraceptive use during the duration of the study.

Exclusion Criteria:

* Allergic to Deoxyribonuclease eye drops or any similar products, or excipients of Deoxyribonuclease eye drops 0.1%.
* Receiving or have received within 30 days any experimental systemic medication.
* Active ocular infection or ocular allergies.
* Any history of eyelid surgery or ocular surgery within the past 3 months.
* Corneal epithelial defect larger than 1 mm2 in either eye.
* The use of topical cyclosporine or corticosteroids within 2 weeks of enrollment
* Have active drug/alcohol dependence or abuse history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-07; Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jain, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Translational Clinic of Corneal Neurobiology laboratory, Illinois Eye and Ear Infirmary, University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Tibrewal S, Sarkar J, Jassim SH, Gandhi S, Sonawane S, Chaudhary S, Byun YS, Ivanir Y, Hallak J, Horner JH, Newcomb M, Jain S. Tear fluid extracellular DNA: diagnostic and therapeutic implications in dry eye disease. Invest Ophthalmol Vis Sci. 2013 Dec 11;54(13):8051-61. doi: 10.1167/iovs.13-12844. PMID 24255046
- [Background] Sonawane S, Khanolkar V, Namavari A, Chaudhary S, Gandhi S, Tibrewal S, Jassim SH, Shaheen B, Hallak J, Horner JH, Newcomb M, Sarkar J, Jain S. Ocular surface extracellular DNA and nuclease activity imbalance: a new paradigm for inflammation in dry eye disease. Invest Ophthalmol Vis Sci. 2012 Dec 17;53(13):8253-63. doi: 10.1167/iovs.12-10430. PMID 23169882
- See also: Principal Investigator description — https://chicago.medicine.uic.edu/directory/name/sandeep-jain-md-jain/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center study was conducted at the Department of Ophthalmology Clinical Trials and Translational Center, the University of Illinois at Chicago (UIC).
Pre-assignment Details: A 2-week washout period was required if topical corticosteroids or topical cyclosporine were discontinued before enrollment.
Period: Overall Study
Arm/Group | DNase | Vehicle
Started | 25 | 22
Completed | 21 | 20
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DNase | Vehicle | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57 [44 to 64] | 55.5 [50.2 to 60.8] | 56 [47 to 62.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47
Diagnosis [Count of Participants; unit: Participants]
  Sjogren's Syndrome | 13 | 12 | 25
  Non-Sjogren's DED | 8 | 6 | 14
  Ocular GVHD | 4 | 4 | 8
OSDI [Median (Inter-Quartile Range); unit: units on a scale] — Ocular Surface Disease Index (OSDI), 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
  units on a scale | 50 [32.5 to 62.5] | 49 [36.6 to 72.9] | 50 [33.65 to 71.335]
Corneal Staining [Median (Inter-Quartile Range); unit: units on a scale] — Corneal staining score as measured by Rose Bengal (RB) dye staining using National Eye Institute (NEI) grading scale. The dye was applied to each eye and a slit lamp was used to observe corneal staining. The NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores with a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with RB dye defined as a score of 0 indicating the best outcome.
  units on a scale
    Oculus Dexter (OD) | 5 [3 to 7] | 5 [4 to 8] | 5 [3 to 6.25]
    Oculus Sinister (OS) | 5 [3 to 6] | 5 [4 to 8] | 5 [4 to 7]
Mucoid Debris Strands [Count of Participants; unit: Participants]
  OD | 20 | 17 | 37
  OS | 16 | 19 | 35
Schirmer I [Median (Inter-Quartile Range); unit: mm] — The Schirmer's I tests consists of a thin strip of filter paper placed in lower conjunctival fornix (between the lower eyelid and ocular surface) for 5 minutes. The length of wetting of the strip is used as a measure of tear production by the eye. A normal level of production is considered to be over 10 millimeters (mm) of tears on the paper. Anything under 10 mm is considered to be an abnormally low level of tear production. A measurement of less than 5 mm is considered severe dry eye.
  mm
    OD | 2 [0 to 4] | 0.75 [0 to 1] | 1 [0 to 2.5]
    OS | 2 [0 to 5] | 0.25 [0 to 1.75] | 1 [0 to 4]
Conjunctival Staining [Median (Inter-Quartile Range); unit: units on a scale] — Conjunctival staining score as measured by Rose Bengal (RB) dye staining using National Eye Institute (NEI) grading scale. The dye was applied to each eye and a slit lamp was used to observe conjunctival staining. The NEI scale relies on a chart that divides the conjunctiva into 2 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores, for a range of 0-6 points. Complete conjunctival staining clearance with RB dye defined as a score of 0 indicating the best outcome.
  units on a scale
    OD | 4.00 [2 to 4] | 4.00 [3 to 6] | 4 [2 to 4.75]
    OS | 4.00 [2 to 4] | 4.00 [2 to 5] | 4 [2 to 4]
Conjunctival Injection [Median (Inter-Quartile Range); unit: units on a scale] — Ocular surface redness (nasal or temporal) will be assessed using the Validated Bulbar Redness grading scale (VBR). VBR consists of 10 images illustrating different degrees of ocular surface redness (OR), ranging from normal to severe, and each image is assigned a value in an order of ascending severity (10-100). Subjects were examined by a slit-lamp and the bulbar conjunctival injection of the subject's eye (nasal and temporal) will be compared to the reference images and graded accordingly.
  units on a scale
    Temporal OD | 40 [30 to 60] | 45 [40 to 60] | 40 [40 to 60]
    Temporal OS | 40 [40 to 60] | 45 [40 to 60] | 40 [40 to 60]
    Nasal OD | 40 [30 to 50] | 40 [40 to 57.5] | 40 [35 to 50]
    Nasal OS | 40 [30 to 50] | 45 [40 to 60] | 40 [30 to 60]
Corneal Filaments [Count of Participants; unit: Participants]
  OD | 0 | 4 | 4
  OS | 1 | 2 | 3
Tolerability [Oculus Uterque (OU)] [Count of Participants; unit: Participants] — To see how subjects react to the study medication, their first dose was given by the investigator at baseline visit in the clinic itself. Afterward, subjects were asked to rate tolerability of the drug on the Visual Analogue Scale (VAS). The VAS is a 100 mm horizontal line with verbal descriptors at either end. The VAS ratings were completed after the administration of the test medication. Subjects placed a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm). Population: Missing data for one patient.
  Participants
    Tolerability (90): number analyzed (Participants) | 25 | 21 | 46
    Tolerability (90) | 2 | 0 | 2
    Tolerability (100): number analyzed (Participants) | 25 | 21 | 46
    Tolerability (100) | 23 | 21 | 44
Intraocular Pressure (IOP) [Median (Inter-Quartile Range); unit: mmHg]
  OD | 17.5 [15 to 20] | 18 [16 to 20] | 18 [15.625 to 20]
  OS | 18.5 [16 to 22] | 18 [15.5 to 20] | 18 [16 to 21]

OUTCOME MEASURES:

1. Primary Outcome: The Change in Corneal Surface Staining as Measured by Rose Bengal Dye Staining
Description: Corneal staining score as measured by Rose Bengal (RB) dye staining using National Eye Institute (NEI) 1995 workshop grading scale. The dye was applied to each eye and a slit lamp was used to observe corneal staining. The NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores, for a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with RB dye defined as a score of 0 indicating the best outcome.
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DNase | Vehicle
Number analyzed (Participants) | 21 | 20
score on a scale
  OD | -1.00 [-3.00 to -1.00] | 0.00 [-0.25 to 1.00]
  OS | -1.00 [-3.00 to -1.00] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: DNase vs Vehicle; Test type: Other; p = 0.001, Kruskal-Wallis

2. Primary Outcome: The Change in the Ocular Surface Disease Index Score
Description: Ocular Surface Disease Index (OSDI), a 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in the past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DNase | Vehicle
Number analyzed (Participants) | 21 | 20
score on a scale
  OD | -20.75 [-37 to -11.80] | -8.43 [-25 to -0.7]
  OS | -20.75 [-37 to -11.80] | -8.43 [-25 to -0.7]
Statistical Analysis 1: Comparison: DNase vs Vehicle; Test type: Other; p = 0.078, Kruskal-Wallis

3. Other Pre Specified Outcome: The Change in Mucoid Debris Strands Between Baseline and 8-weeks
Description: The presence of mucoid debris/strands over the ocular surface was assessed and the amount graded as the absence of mucoid debris (0) or presence of mucoid debris (1+, 2+ or 3+) with a bigger number indicating greater presence of mucoid debris with "3+" implying presence of the highest amount of mucoid debris and indicating the worst outcome.
Time Frame: Between baseline and 8-weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DNase | Vehicle
Number analyzed (Participants) | 21 | 20
score on a scale
  OD | -1.00 [-2.00 to 0.00] | 0.00 [0.00 to 1.00]
  OS | 0.00 [-1.00 to 0.00] | 0.00 [0.00 to 0.25]
Statistical Analysis 1: Comparison: DNase vs Vehicle; Test type: Other; p < 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Between baseline and 8-weeks of treatment.
Arm/Group | DNase | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 9/25 | 12/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DNase (N=25) | Vehicle (N=21)
Grittines (Eye disorders) | 4 | 2
Blurred Vision (Eye disorders) | 3 | 3
Burning (Eye disorders) | 5 | 2
Light Sensitivity (Eye disorders) | 1 | 1
Itching (Eye disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
Outcomes of this clinical trial shouldn't be over-interpreted for benefit. Accurate assessment of therapeutic implications of DNase eye drops will only be possible after adequately powered definitive pivotal trials. Small sample size is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02193490/Prot_SAP_000.pdf